CLINICAL TRIAL: NCT03975647
Title: Randomized, Double-blind, Phase 3 Study of Tucatinib or Placebo in Combination With Ado-trastuzumab Emtansine (T-DM1) for Subjects With Unresectable Locally-advanced or Metastatic HER2+ Breast Cancer (HER2CLIMB-02)
Brief Title: A Study of Tucatinib vs. Placebo in Combination With Ado-trastuzumab Emtansine (T-DM1) for Patients With Advanced or Metastatic HER2+ Breast Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Seagen, a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SGNTUC-016; C4251001 (Other: Alias Study Number); 2024-514733-38-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2019-06-04; First posted 2019-06-05 (Actual); Results first posted 2024-07-30 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: HER2-positive Breast Cancer
Keywords: Seattle Genetics; Seagen
MeSH Terms: interventions — tucatinib; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tucatinib + T-DM1 (Experimental): Tucatinib + T-DM1
  Interventions: Drug: tucatinib; Drug: T-DM1
- Placebo + T-DM1 (Active Comparator): Placebo + T-DM1
  Interventions: Drug: placebo; Drug: T-DM1

INTERVENTIONS:
Drug: tucatinib — 300mg given twice per day by mouth (orally)
  Other Names: ONT-380
  Arms: Tucatinib + T-DM1
Drug: placebo — Given twice per day orally
  Arms: Placebo + T-DM1
Drug: T-DM1 — 3.6 mg/kg given into the vein (IV; intravenously) every 21 days
  Other Names: Kadcyla

SUMMARY:
This study is being done to see if tucatinib with ado-trastuzumab emtansine (T-DM1) works better than T-DM1 alone to help patients who have a specific type of breast cancer called HER2 positive breast carcinoma. The breast cancer in this study is either metastatic (spread into other parts of the body) or cannot be removed completely with surgery.

Patients in this study will be randomly assigned to get either tucatinib or placebo (a pill with no medicine). This is a blinded study, so neither patients nor their doctors will know whether a patient gets tucatinib or placebo. All patients in the study will get T-DM1, a drug that is often used to treat this cancer.

Each treatment cycle lasts 21 days. Patients will swallow tucatinib pills or placebo pills two times every day. Patients will get T-DM1 injections from the study site staff on the first day of every cycle.

DETAILED DESCRIPTION:
This study is designed to evaluate the efficacy and safety of tucatinib in combination with T-DM1 in participants with unresectable locally-advanced or metastatic HER2+ breast cancer who have had prior treatment with a taxane and trastuzumab in any setting. Prior pertuzumab treatment is permitted, but not required. Participants will be randomized in a 1:1 manner to receive 21-day cycles of either tucatinib or placebo in combination with T-DM1.

While on study treatment, participants will be assessed for progression every 6 weeks for the first 24 weeks, and every 9 weeks thereafter, irrespective of dose holds or interruptions. Study treatment will continue until unacceptable toxicity, disease progression, withdrawal of consent, or study closure. After completion of study treatment and after occurrence of disease progression, participants in both arms of the study will continue to be followed for survival until study closure or withdrawal of consent.

ELIGIBILITY:
* Inclusion Criteria:

  * Histologically confirmed HER2+ breast carcinoma as determined by a sponsor-designated central laboratory
  * History of prior treatment with a taxane and trastuzumab in any setting, separately or in combination
  * Have progression of unresectable locally advanced/metastatic breast cancer after last systemic therapy, or be intolerant of last systemic therapy
  * Measurable or non-measurable disease assessable by RECIST v1.1
  * ECOG performance status score of 0 or 1
  * CNS Inclusion - Based on screening contrast brain magnetic resonance imaging (MRI), participants must have at least one of the following:

    (a) No evidence of brain metastases

    (b) Untreated brain metastases not needing immediate local therapy

    (c) Previously treated brain metastases
    1. Brain metastases previously treated with local therapy may either be stable since treatment or may have progressed since prior local CNS therapy, provided that there is no clinical indication for immediate re-treatment with local therapy
    2. Participants treated with CNS local therapy for newly identified lesions or previously treated and progressing lesions may be eligible to enroll if all of the following criteria are met:

       (i) Time since SRS is at least 7 days prior to first dose of study treatment, time since WBRT is at least 14 days prior to first dose, or time since surgical resection is at least 28 days.

       (ii) Other sites of evaluable disease are present
    3. Relevant records of any CNS treatment must be available to allow for classification of target and non-target lesions
* Exclusion Criteria:

  * Prior treatment with tucatinib, afatinib, trastuzumab deruxtecan (DS-8201a), or any other investigational anti-HER2, anti-EGFR, or HER2 TKI agent. Prior treatment with lapatinib or neratinib within 12 months of starting study treatment (except in cases where they were given for ≤21 days and was discontinued for reasons other than disease progression or severe toxicity). Prior treatment with pyrotinib for recurrent of mBC (except in cases where pyrotinib was given for ≤21 days and was discontinued for reasons other than disease progression or severe toxicity).
  * CNS Exclusion - Based on screening contrast brain magnetic resonance imaging (MRI), participants must not have any of the following:

    1. Any untreated brain lesions >2 cm in size
    2. Ongoing use of corticosteroids for control of symptoms of brain metastases at a total daily dose of >2 mg of dexamethasone (or equivalent).
    3. Any brain lesion thought to require immediate local therapy
    4. Known or concurrent leptomeningeal disease as documented by the investigator
    5. Poorly controlled generalized or complex partial seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 466 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2029-03-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (473):
- United States (303):
  - University of South Alabama Health Children's and Women's Hospital, Mobile, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - University of South Alabama Health University Hospital, Mobile, Alabama
  - Banner Gateway Medical Center, Gilbert, Arizona
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Western Regional Medical Center, LLC, Goodyear, Arizona
  - Arizona Oncology Associates, PC - HOPE., Tucson, Arizona
  - Arizona Oncology Associates, PC - HOPE, Tucson, Arizona
  - UCLA Hematology/Oncology - Alhambra, Alhambra, California
  - Kaiser Permanente Medical Center Lab Drawing Station, Antioch, California
  - UCLA Hematology/Oncology- Beverly Hills, Beverly Hills, California
  - UC Irvine Health Cancer Center - Newport, Costa Mesa, California
  - City of Hope Investigational Drug Services (IDS), Duarte, California
  - City of Hope(City of Hope National Medical Center,City of Hope Medical Center), Duarte, California
  - Kaiser Permanente Medical Center (Radiology), Dublin, California
  - UCLA Hematology/Oncology - Encino, Encino, California
  - Kaiser Permanente Medical Center Lab Drawing Station, Fairfield, California
  - Kaiser Permanente Medical Center Lab Drawing Station, Gilroy, California
  - UCLA Hematology/Oncology- Irvine, Irvine, California
  - Drug Management Only: UCLA West Medical Pharmacy, Attn: Steven L Wong, Pharm.D., Los Angeles, California
  - Regulatory Management only: TRIO-US Central Administration, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UCLA Hematology/Oncology, Los Angeles, California
  - UCLA West Medical Pharmacy, Los Angeles, California
  - Kaiser Permanente Medical Center Lab Drawing Station, Martinez, California
  - Kaiser Permanente Medical Center Lab Drawing Station, Milpitas, California
  - Kaiser Permanente Medical Center Lab Drawing Station, Modesto, California
  - Kaiser Permanente Medical Center Lab Drawing Station, Mountain View, California
  - Kaiser Permanente Medical Center Lab Drawing Station, Napa, California
  - Kaiser Permanente Medical Center (clinic+DSL), Oakland, California
  - Kaiser Permanente Medical Center (Radiology), Oakland, California
  - Chao Family Comprehensive Cancer Center University of California Irvine, Orange, California
  - UC Irvine Medical Center Attn: Trisha Maris, Orange, California
  - UCI Medical Center - Chao Family Comprehensive Cancer Center, Orange, California
  - Kaiser Permanente Medical Center Lab Drawing Station, Pleasanton, California
  - UCLA Hematology/Oncology - Porter Ranch, Porter Ranch, California
  - Kaiser Permanente Medical Center Lab Drawing Station, Redwood City, California
  - Kaiser Permanente Medical Center (clinic+DSL), Roseville, California
  - Kaiser Permanente Sacramento J Street Medical Center (clinic+DSL+Lab Drawing Station), Sacramento, California
  - University of California Davis Medical Center, Sacramento, California
  - University of California Davis, Sacramento, California
  - Kaiser Permanente Medical Center (Radiology), Sacramento, California
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - Kaiser Permanente Medical Center (clinic+DSL), San Francisco, California
  - University of California, San Francisco (UCSF) Helen Diller Family Comprehensive Cancer Center., San Francisco, California
  - Kaiser Permanente Mission Bay Medical Center Lab Drawing Station, San Francisco, California
  - Kaiser Permanente Medical Center Lab Drawing Station, San Jose, California
  - Kaiser Permanente Medical Center (clinic+DSL), San Jose, California
  - Kaiser Permanente Medical Center (clinic+DSL), San Leandro, California
  - UCLA Hematology/Oncology - San Luis Obispo, San Luis Obispo, California
  - Kaiser Permanente Medical Center (clinic+DSL), Santa Clara, California
  - UCLA Hematology/Oncology - Santa Monica, Santa Monica, California
  - UCLA Hematology/Oncology Parkside, Santa Monica, California
  - Kaiser Permanente Medical Center (clinic+DSL), South San Francisco, California
  - Torrance Memorial Physician Network - Cancer Care, Torrance, California
  - Torrance Memorial Physician Network-Cancer Care, Torrance, California
  - UCLA Torrance Oncology, Torrance, California
  - UCLA Hematology/Oncology - Santa Clarita, Valencia, California
  - Kaiser Permanente Medical Center (clinic+DSL), Vallejo, California
  - UCLA Hematology/Oncology - Ventura, Ventura, California
  - Kaiser Permanente Medical Center (clinic+DSL), Walnut Creek, California
  - Rocky Mountain Cancer Centers, LLP, Aurora, Colorado
  - Clinical and Translational Research Center (CTRC), Aurora, Colorado
  - University of Colorado Hospital - Anschutz Cancer Pavilion(ACP), Aurora, Colorado
  - University of Colorado Hospital - Anschutz Inpatient Pavilion (AIP), Aurora, Colorado
  - University of Colorado Hospital - Anschutz Outpatient Pavilion (AOP), Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Rocky Mountain Cancer Centers, LLP, Boulder, Colorado
  - Rocky Mountain Cancer Centers, LLP, Centennial, Colorado
  - Rocky Mountain Cancer Centers, LLP, Colorado Springs, Colorado
  - UCH-MHS Memorial Hospital Central, Colorado Springs, Colorado
  - Printers Park Medical Plaza, Colorado Springs, Colorado
  - Briargate Medical Campus, Colorado Springs, Colorado
  - UCH-MHS Memorial Hospital North, Colorado Springs, Colorado
  - UCHealth Cherry Creek Medical Center, Denver, Colorado
  - UCHealth IDS Research Pharmacy - Cherry Creek, Denver, Colorado
  - Cancer Centers of Colorado at Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers, LLP, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care & Hematology - Fort Collins, Fort Collins, Colorado
  - Cancer Care & Hematology - Greeley, Greeley, Colorado
  - SCL Health Good Samaritan Medical Center Cancer Centers of Colorado, Lafayette, Colorado
  - SCL Health Good Samaritan Medical Center, Lafayette, Colorado
  - Rocky Mountain Cancer Centers, LLP, Lakewood, Colorado
  - Rocky Mountain Cancer Centers, LLP, Littleton, Colorado
  - Rocky Mountain Cancer Centre, LLP, Lone Tree, Colorado
  - Cancer Care & Hematology - Loveland, Loveland, Colorado
  - Rocky Mountain Cancer Centers, LLP, Thornton, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Washington Cancer Institute at MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Florida Cancer Specialists, Altamonte Springs, Florida
  - Florida Cancer Specialists, Bonita Springs, Florida
  - Florida Cancer Specialists, Brandon, Florida
  - Florida Cancer Specialists, Cape Coral, Florida
  - Florida Cancer Specialists, Clearwater, Florida
  - Sylvester Comprehensive Cancer Center - The Lennar Foundation Medical Center, Coral Gables, Florida
  - Florida Cancer Specialists., Daytona Beach, Florida
  - Sylvester Comprehensive Cancer Center- Deerfield Beach, Deerfield Beach, Florida
  - Florida Cancer Specialists - South Region, Fort Myers, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Specialists, Gainesville, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Florida Cancer Specialists, Largo, Florida
  - Florida Cancer Specialists, Lecanto, Florida
  - Bascom Palmer Eye Institute, Miami, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Miami Cancer Institute at Baptist Health, Inc., Miami, Florida
  - Sylvester Comprehensive Cancer Center Kendall, Miami, Florida
  - Florida Cancer Specialists, Naples, Florida
  - Florida Cancer Specialists, Ocala, Florida
  - AdventHealth Orlando, Orlando, Florida
  - AdventHealth Hematology and Oncology, Orlando, Florida
  - AdventHealth Medical Group Orlando, Orlando, Florida
  - AdventHealth Orlando Infusion Center, Orlando, Florida
  - AdventHealth Orlando, Investigational Drug Services, Orlando, Florida
  - Florida Cancer Specialists, Orlando, Florida
  - Orlando Health, Inc. TRIO, Orlando, Florida
  - Sylvester Comprehensive Cancer Center Plantation, Plantation, Florida
  - Florida Cancer Specialists, Port Charlotte, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - Florida Cancer Specialists - North Region, St. Petersburg, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Florida Cancer Specialists., Stuart, Florida
  - Florida Cancer Specialists, Tampa, Florida
  - Moffitt Cancer Center, Richard M, Schulze Family Foundation Outpatient Center at McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Moffitt McKinley Hospital, Tampa, Florida
  - Florida Cancer Specialists, Tavares, Florida
  - Florida Cancer Specialists, The Villages, Florida
  - Florida Cancer Specialists, Trinity, Florida
  - Florida Cancer Specialists., Vero Beach, Florida
  - Florida Cancer Specialists., Wellington, Florida
  - Florida Cancer Specialists., West Palm Beach, Florida
  - Northside Hospital, Inc. - GCS/ Athens, Athens, Georgia
  - Winship Cancer Institute, Emory University., Atlanta, Georgia
  - Atlanta Cancer Care - Atlanta, Atlanta, Georgia
  - Northside Hospital, Inc. - Central Research Department, Atlanta, Georgia
  - Northside Hospital, Inc. - GCS/Northside, Atlanta, Georgia
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - Northside Hospital, Inc. - GCS/Blairsville, Blairsville, Georgia
  - Northside Hospital, Inc. - GCS/Canton, Canton, Georgia
  - Atlanta Cancer Care - Cumming, Cumming, Georgia
  - Northside Hospital, Inc. - GCS/Macon, Macon, Georgia
  - Northside Hospital, Inc. - GCS/Kennestone, Marietta, Georgia
  - Hawai'i Pacific Health Research Institute - Administrative Site, Honolulu, Hawaii
  - Kaiser Permanente Hawaii., Honolulu, Hawaii
  - Kaiser Permanente Hawaii, Honolulu, Hawaii
  - Kapi'olani Medical Center for Women and Children, Honolulu, Hawaii
  - Kapi'olani Women's Center, Honolulu, Hawaii
  - Illinois CancerCare- Bloomington, Bloomington, Illinois
  - Rush University Medical Center, Professional Office Building Infusion Pharmacy, Chicago, Illinois
  - Rush University Medical Center., Chicago, Illinois
  - University of Chicago Medical Center, CCD- Investigational Drug Service Pharmacy, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Illinois CancerCare - Galesburg, Galesburg, Illinois
  - University of Chicago Comprehensive Cancer Center at Silver Cross Hospital, New Lenox, Illinois
  - Orland Park - University of Chicago Center for Advanced Care, Orland Park, Illinois
  - Illinois CancerCare- Pekin, Pekin, Illinois
  - Illinois CancerCare, P.C., Peoria, Illinois
  - Illinois CancerCare- Peru, Peru, Illinois
  - Ft Wayne Medical Oncology and Hematology, Inc TRIO, Fort Wayne, Indiana
  - The University of Kansas Cancer Center - West, Kansas City, Kansas
  - MidAmerica Division, Inc. c/o Menorah Medical Center, Overland Park, Kansas
  - The University of Kansas Cancer Center - Overland Park, Overland Park, Kansas
  - The University of Kansas Cancer Center - Indian Creek Campus, Overland Park, Kansas
  - The University of Kansas Cancer Center Breast Surgery Center - Indian Creek Campus, Overland Park, Kansas
  - The University of Kansas Cancer Center, Investigational Drug Services, Westwood, Kansas
  - The University of Kansas Cancer Center, Westwood, Kansas
  - CHI Saint Joseph Cancer Care, Lexington, Kentucky
  - Saint Joseph Health Infusion Services, Lexington, Kentucky
  - University of Maryland, Greenebaum Comprehensive Cancer Center., Baltimore, Maryland
  - Mercy Medical Center -Weinberg Center, Baltimore, Maryland
  - Mercy Medical Center., Baltimore, Maryland
  - Maryland Oncology Hematology, P.A, Bethesda, Maryland
  - Maryland Oncology Hematology, P.A, Brandywine, Maryland
  - Maryland Oncology Hematology, P.A, Columbia, Maryland
  - Maryland Oncology Hematology, P.A, Frederick, Maryland
  - Maryland Oncology Hematology, P.A, Largo, Maryland
  - Maryland Oncology Hematology, P.A, Rockville, Maryland
  - Maryland Oncology Hematology, P.A, Silver Spring, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana Farber Cancer Institute- Chestnut Hill, Newton, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Brighton Center for Specialty Care, Brighton, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Minnesota Oncology Hematology, P.A., Edina, Minnesota
  - Siteman Cancer Center - St Peters, City of Saint Peters, Missouri
  - Siteman Cancer Center - West County, Creve Coeur, Missouri
  - Siteman Cancer Center - North County, Florissant, Missouri
  - MidAmerica Division, Inc. c/o Centerpoint Medical Center, Independence, Missouri
  - Saint Luke's Cancer institute, Kansas City, Missouri
  - The University of Kansas Cancer Center, Kansas City, Missouri
  - MidAmerica Division, Inc., c/o Research Medical Center, Kansas City, Missouri
  - The University of Kansas Cancer Center -North, Kansas City, Missouri
  - The University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine - Siteman Cancer Center., St Louis, Missouri
  - Washington University School of Medicine - St. Louis, St Louis, Missouri
  - Siteman Cancer Center - South County, St Louis, Missouri
  - St. Vincent Healthcare, Billings, Montana
  - St. Vincent - Frontier Cancer Center, Billings, Montana
  - Saint Luke's Hospital Investigational Pharmacy, Ronan, Montana
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists, Omaha, Nebraska
  - West Omaha Imaging, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada Research Department, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Summit Medical Group, Berkeley Heights, New Jersey
  - Summit Medical Group, Florham Park, New Jersey
  - Cooperman Barnabas Medical Center, Livingston, New Jersey
  - New York Oncology Hematology, P.C., Albany, New York
  - Stony Brook Advanced Imaging, Stony Brook, New York
  - Stony Brook Cancer Center, Stony Brook, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Carolinas Medical Center (biopsy only), Charlotte, North Carolina
  - Charlotte Radiology Medical Center Plaza Breast Center (biopsy only), Charlotte, North Carolina
  - Carolinas Medical Center Investigational Drug Services, Charlotte, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - Carolinas Medical Center - Mercy (biopsy only), Charlotte, North Carolina
  - Atrium Health Pineville (biopsy only), Charlotte, North Carolina
  - Levine Cancer Institute-Pineville, Charlotte, North Carolina
  - Atrium Health University City (biopsy only), Charlotte, North Carolina
  - Atrium Health Cabarrus (biopsy only), Concord, North Carolina
  - Levine Cancer Institute Concord, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Atrium Health Union (biopsy only), Monroe, North Carolina
  - OHSU Knight Cancer Institute, Beaverton, Beaverton, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - OHSU Knight Cancer Institute, Gresham, Gresham, Oregon
  - OHSU Knight Cancer Institute, Northwest Portland, Portland, Oregon
  - Northwest Cancer Specialists P.C., Portland, Oregon
  - Providence Cancer Institute Franz Clinic, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - OHSU Knight Cancer Institute, East Portland, Portland, Oregon
  - OHSU Center for Health and Healing 2, Portland, Oregon
  - OHSU Center for Health and Healing, Portland, Oregon
  - OHSU Research Pharmacy Services, Portland, Oregon
  - Oregon Health And Science University, Portland, Oregon
  - Northwest Cancer Specialists, P.C., Tigard, Oregon
  - OHSU Knight Cancer Institute, Tualatin, Tualatin, Oregon
  - Hospital of the University of Pennsylvania, Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Tennessee Oncology PLLC, Dickson, Tennessee
  - Tennessee Oncology PLLC, Franklin, Tennessee
  - Tennessee Oncology PLLC, Gallatin, Tennessee
  - Tennessee Oncology PLLC, Hendersonville, Tennessee
  - Tennessee Oncology PLLC, Hermitage, Tennessee
  - Brig Center for Cancer Care and Survivorship, Knoxville, Tennessee
  - Tennessee Oncology PLLC, Lebanon, Tennessee
  - Tennessee Oncology PLLC, Murfreesboro, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - The Sarah Cannon Research Institute, Nashville, Tennessee
  - Tennessee Oncology PLLC, Shelbyville, Tennessee
  - Tennessee Oncology PLLC, Smyrna, Tennessee
  - Texas Oncology - West Texas, Amarillo, Texas
  - The Center for Cancer and Blood Disorders, Arlington, Texas
  - Texas Oncology - Austin, Austin, Texas
  - Texas Oncology - DFWW, Bedford, Texas
  - Texas Oncology - DFW, Bedford, Texas
  - The Center for Cancer and Blood Disorders, Burleson, Texas
  - Texas Oncology - DFW, Dallas, Texas
  - Parkland Health and Hospital System, Dallas, Texas
  - Texas Oncology - DFWW, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - UT Southwestern Medical Center - Simmons Cancer Center Pharmacy, Dallas, Texas
  - UT Southwestern Medical Center - Simmons Cancer Center, Dallas, Texas
  - UT Southwestern University Hospital - William P. Clements, Jr, Dallas, Texas
  - UT Southwestern University Hospital - Zale Lipshy, Dallas, Texas
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - UT Southwestern Medical Center - d/b/a Moncrief Cancer Institute - Ft. Worth - Pharmacy, Fort Worth, Texas
  - UT Southwestern Medical Center d/b/a Moncrief Cancer Institute - Ft. Worth, Fort Worth, Texas
  - Oncology Consultants, P.A., Houston, Texas
  - Texas Oncology - Gulf Coast, Houston, Texas
  - Baylor College of Medicine Medical center, Houston, Texas
  - Baylor St. Luke's Medical Center, Houston, Texas
  - Harris Health System - Ben Taub General Hospital, Houston, Texas
  - Harris Health System - Smith Clinic, Houston, Texas
  - Texas Oncology - San Antonio, New Braunfels, Texas
  - UT Southwestern Medical Center - Clinical Center Richardson/Plano - Pharmacy, Richardson, Texas
  - UT Southwestern Medical Center - Clinical Center Richardson/Plano, Richardson, Texas
  - Texas Oncology-San Antonio, San Antonio, Texas
  - The Center for Cancer and Blood Disorders, Weatherford, Texas
  - University of Utah, Farmington Health Center, Farmington, Utah
  - University of Utah, Sugar House Health Center, Salt Lake City, Utah
  - University of Utah, Huntsman Cancer Hospital, Salt Lake City, Utah
  - University of Utah, Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Utah, South Jordan Health Center, South Jordan, Utah
  - Virginia Cancer Specialists, PC, Alexandria, Virginia
  - Virginia Cancer Specialists, PC, Arlington, Virginia
  - Oncology & Hematology Associates of Southwest Virginia,Inc.DBA Blue Ridge Cancer Care, Blacksburg, Virginia
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Cancer Specialists, PC, Gainesville, Virginia
  - Virginia Cancer Specialists, PC, Leesburg, Virginia
  - Oncology and Hematology Associates of Southwest Virginia Inc, Low Moor, Virginia
  - Oncology & Hematology Associates of Southwest Virginia,Inc.DBA Blue Ridge Cancer Care, Roanoke, Virginia
  - Oncology & Hematology Associates of Southwest Virginia,Inc.DBA Blue Ridge Cancer Care, Salem, Virginia
  - Oncology and Hematology Associates of Southwest Virginia Inc, Wytheville, Virginia
  - Swedish Cancer Institute - Edmonds Campus, Edmonds, Washington
  - Swedish Cancer Institute - Issaquah Campus, Issaquah, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
  - Northwest Cancer Specialists P.C., Vancouver, Washington
- Australia (9):
  - Patricia Ritchie Centre for Cancer Care and Research Mater Hospital Sydney, North Sydney, New South Wales
  - The Crown Princess Mary Cancer Centre, Westmead Hospital, Westmead, New South Wales
  - Austin Health, Heidelberg, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
  - Epic Pharmacy Hollywood, Nedlands, Western Australia
  - Hollywood Private Hospital, Nedlands, Western Australia
  - Starcevich Day Clinic, Hollywood Private Hospital, Nedlands, Western Australia
  - Breast Cancer Research Centre - WA, Nedlands
- Austria (4):
  - Universitatsklinik Innsbruck fur Gynakologie und Geburtshilfe BrustGesundheitzentrum, Innsbruck
  - CT/MRIfacility:Diagnosezentrum Urania, Vienna
  - Klinik Ottakring., Vienna
  - Wilhelminen Krebsforschung GmbH, Vienna
- Belgium (8):
  - Institut Jules Bordet, Anderlecht, Bruxelles-capitale, Région de
  - Clinical Trails Conduct Unit(CTCU) Institut Jules Bordet, Brussels
  - GHdC, Charleroi
  - University Hospital Antwerp, Edegem
  - AZ Groeninge, Kortrijk
  - UZ Leuven, Leuven
  - CHU de Liege, Liège
  - CHU UCL Site Sainte Elisabeth, Namur
- Canada (6):
  - Cross Cancer Institute, Edmonton, Alberta
  - London Regional Cancer Program, London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Motreal (CHUM), Montreal, Quebec
  - CHU de Québec-Université Laval, St-Sacrement Hospital, Québec
- China (24):
  - Maternal and child Health Hospital of Guangdong Province, Guangzhou, Guangdong
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital., Changsha, Hu'nan
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Nanjing Drum Tower Hospital , The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Nanchang Third Hospital, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - Shengjing Hospital Of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Xi'an International Medical Center Hospital, Xi’an, Shanxi
  - Zigong First People's Hospital, Zigong, Sichuan
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Beijing Hospital, Beijing
  - Cancer Hospital Chinese Academy of medical sciences, Beijing
  - Peking University People's Hospital, Beijing
  - Zhejiang Cancer Hospital, Hangzhou
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning
  - Tianjin Cancer Hospital, Tianjin
- Denmark (8):
  - Blandecentralen Odense Universitetshospital, Odense C, Other
  - Onkologisk Afdeling R, Odense Universitetshospital, Odense C, Other
  - Pharmacy., Vejle, Other
  - Herlev og Gentofte Hospital, Herlev
  - Pharmacy : Region Hovedstadens Apotek-KFS Serviceproduktion - Cytostatikaenheden, Herlev
  - Radiology: Herlev - og Gentofte Hospital - Radiologisk afdeling, Herlev
  - Radiology., Vejle
  - Vejle Sygehus, Vejle
- France (32):
  - University Hospital of Besancon, Besançon, Other
  - Service de Pharmacie Centre Francois Baclesse, Caen, Other
  - Service de radiologie Centre Francois Baclesse, Caen, Other
  - Department de Radiodiagnostic Centre GF Leclerc, Dijon, Other
  - Service Pharmacie Centre GF Leclerc, Dijon, Other
  - Centre Leon Berard - Centre regional de lutte contre le cancer Rhone-Alpes, Lyon, Other
  - Departement de radiologie Hopital Bretonneau - CHRU de Tours, Tours, Other
  - Hopital Bretonneau CHRU de Tours, Tours, Other
  - Pharmacie Hopital Bretonneau - CHRU de Tours, Tours, Other
  - Departement de radiologie Clinique Victor Hugo, Le Mans, Sarthe
  - CHRU Besancon Service Radiologie, Besançon
  - CHRU Besancon, Besançon
  - Dimeo lmagerie Medicale Polyclinique - Besancon, Besançon
  - CHRU Morvan Pharmacie des essais cliniques, Brest
  - CHRU Morvan Unité de recherche clinique en cancérologie, Brest
  - Centre Francois Baclesse, Caen
  - Centre GF Leclerc, Dijon
  - Clinique du mail, Grenoble
  - Clinique Victor Hugo Centre de Cancerologie de la Sarthe, Le Mans
  - Centre Leon Berard Departement de Medecine, Lyon
  - Departement de radiologie Centre Leon Berard, Lyon
  - Pharmacie - Secteur essais Cliniques Centre Leon Berard, Lyon
  - Pharmacie des essais cliniques -lnstitut Paoli calmettes, Marseille
  - lnstitut Paoli Calmettes, Departement ONCOLOGIE MEDICALE, Marseille
  - Groupement hospitalier Portes de Provence Quartier Beausseret, Montélimar
  - Departement d'imagerie medicale Institut Curie - Site Paris, Paris
  - lnstitut Curie- Site Paris, Paris
  - Centre Paul Strauss - pharmacie, Strasbourg
  - lnstitut de cancerologie Strasbourg Europe, Strasbourg
  - IUCT-O, Toulouse
  - lnstitut Claudius Regaud - IUCT-O, Toulouse
  - Hopital Nord Franche-Comte Pole imagerie radiologie, Trévenans
- Germany (5):
  - Universitatsmedizin Mainz, Mainz, Other
  - Universitaetsklinikum Schieswig-Holstein, Campus Kiel, Klinik f. Gynaekologie und Geburtshilfe, Kiel
  - InVO-lnstitut für Versorgungsforschung in der Onkologie GbR, Koblenz
  - Klinikum rechts der Isar, Klinik und Poliklinik fur Frauenheikunde, München
  - Sana Klinikum Offenbach GmbH Zentralinstitut fur Diagnostische und Interventionelle Radiologie, Offenbach/ Main
- Israel (3):
  - Oncology Institute, Meir Medical Center, Kfar Saba
  - Institute of Oncology - Davidoff Center, Rabin Medical Center, Beilinson Hospital, Petah Tikva
  - Oncology Institute, Kaplan Medical Center, Rehovot
- Italy (10):
  - A.O.U. Ospedali Riuniti di Ancona., Torrette, Ancona
  - Azienda Ospedaliero Universitaria di Bologna - IRCCS, Bologna, Emilia-Romagna
  - Azienda Ospedaliero-Universitaria di Bologna Policlinico S. Orsola-Malpighi, Bologna, Emilia-Romagna
  - Fondazione Policlinico Gemelli IRCCS, Rome, Lazio
  - AUSL della Romagna. P.O. Ospedale degli lnfermi. U.O. di Oncologia., Faenza, Ravenna
  - AUSL della Romagna. P.O. Ospedale di Lugo Umberto I. U.O. di Oncologia., Lugo, Ravenna
  - AUSL della Romagna. P.O. Ospedale Cervesi. U.O. di Oncologia., Cattolica, Rimini
  - lstituto Europeo di Oncologia, Milan
  - AUSL della Romagna. P.O. Ospedale Santa Maria delle Croci. U.O. di Oncologia., Ravenna
  - AUSL della Romagna P.O. Ospedale Infermi U.O. di Oncologia, Rimini
- Japan (23):
  - Nagoya Radiological Diagnosis Foundation, East Nagoya Imaging Diagnosis Center, Nagoya, Aichi-ken
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East., Kashiwa, Chiba
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima, Chūgoku
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - National Hospital Organization Kyushu Cancer Center., Fukuoka, Fukuoka
  - National Hospital Organization Hokkaido Cancer Center., Sapporo, Hokkaido
  - Hyogo college of medicine hospital, Nishinomiya, Hyōgo
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Hakuaikai Medical Corporation Sagara Hospital, Kagoshima, Kagoshima-ken
  - Hakuaikai Medical Corporation Sagara Perth Street Clinic, Kagoshima, Kagoshima-ken
  - Koyasu Neurosurgical Clinic, Yokohama, Kanagawa
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Morinomiya Hospital, Osaka, Osaka
  - Saitama Cancer Center, Breast Oncology, Kitaadachi-gun, Saitama
  - Shizuoka Cancer Center, Nagaizumi-cho, Shizuoka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Chiba Cancer Center, Chiba
  - Advanced Imaging Center, Ibaraki
  - Kumamoto Shinto General Hospital, Kumamoto
  - National Hospital Organization Osaka National Hospital, Osaka
  - Osaka Prefectural Hospital Organization Osaka International Cancer Institute, Osaka
  - The Cancer Institute Hospital of JFCR, Tokyo
- Netherlands (3):
  - Amphia Ziekenhuis, Breda
  - Martini Ziekenhuis, Groningen
  - Erasmus Medisch Centrum Daniel Den Hoed, Rotterdam
- Singapore (2):
  - National Cancer Centre Singapore, Singapore, Other
  - National University Hospital, Singapore
- South Korea (7):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - National Cancer Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (14):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Quiron Barcelona, Barcelona, Other
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa CRUZ DE Tenerife
  - Vall d'Hebron University Hospital, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Clinica Nuestra Senora del Rosario, Madrid
  - Hospital Ruber Internacional, Madrid
  - Hospital Universitario Clinico San Carlos, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Moises Broggi- ICO, Sant Joan Despí
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Quirón Zaragoza, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Onkologkliniken, KPE, Malpunkt K,, J0nkoping
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital Winterthur Onkologie, Winterthur
- Taiwan (2):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- United Kingdom (6):
  - The Royal Cornwall Hospital, Truro, Cornwall
  - "Edinburgh Cancer Centre, Western General Hospital,", Edinburgh, Scotland
  - University Hospitals Birmingham NHS Foundation Trust Queen Elizabeth Hospital, Birmingham
  - The Royal Marsden NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - The Royal Marsden NHS Foundation Trust, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Hurvitz SA, Loi S, O'Shaughnessy J, Okines AFC, Tolaney SM, Sohn J, Saura C, Zhu X, Cameron D, Bachelot T, Hamilton E, Curigliano G, Wolff AC, Harbeck N, Masuda N, Vahdat L, Zaman K, Valdes-Albini F, Block M, Pluard T, Tan TJ, Gawryletz C, Chan A, Bedard PL, Yerushalmi R, Xu B, Schmitt M, Xie D, Borges VF; HER2CLIMB-02 study investigators. Tucatinib and trastuzumab emtansine for patients with previously treated HER2-positive locally advanced and metastatic breast cancer: primary analysis of the randomized phase III trial HER2CLIMB-02. Ann Oncol. 2025 Nov 17:S0923-7534(25)06263-5. doi: 10.1016/j.annonc.2025.11.005. Online ahead of print. PMID 41260264
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=SGNTUC-016

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants diagnosed with locally advanced (LA) or metastatic human epidermal growth factor receptor 2 positive (HER2+) breast cancer who received prior treatment with a taxane and trastuzumab in any setting, were evaluated for efficacy and safety of tucatinib in combination with ado-trastuzumab emtansine (T-DM1) in this study.
Pre-assignment Details: A total of 618 participants were screened of which 152 failed screening and 466 participants were enrolled in the study.
Groups:
- Tucatinib+ Ado-trastuzumab Emtansine: Participants with HER2+ LA/mBC were treated with tucatinib 300 mg orally twice a day (BID) and T-DM1 3.6 mg/kg IV every 21 days in each 21-day cycle. Participants received treatment until unacceptable toxicity, disease progression, withdrawal of consent, or study closure.
- Placebo+ Ado-trastuzumab Emtansine: Participants with HER2+ LA/mBC were treated with placebo orally BID, and T-DM1 3.6 mg/kg IV every 21 days in each 21-day cycle. Participants received treatment until unacceptable toxicity, disease progression, withdrawal of consent, or study closure.
Period: Overall Study
Arm/Group | Tucatinib+ Ado-trastuzumab Emtansine | Placebo+ Ado-trastuzumab Emtansine
Started | 231 | 235
Intent-to-Treat (ITT) Analysis Set | 228 | 235
Completed | 151 | 159
Not Completed | 80 | 76
Not completed — Death | 71 | 63
Not completed — Lost to Follow-up | 2 | 2
Not completed — Subject withdrawal of consent | 7 | 11

BASELINE CHARACTERISTICS:
Population: The ITT analysis set included all participants who were randomized on or before the date of last patient in (LPI) in the global study.
Groups:
- Tucatinib+ Ado-trastuzumab Emtansine: Participants with HER2+ LA/mBC were treated with tucatinib 300 mg orally BID and T-DM1 3.6 mg/kg IV every 21 days in each 21-day cycle. Participants received treatment until unacceptable toxicity, disease progression, withdrawal of consent, or study closure.
- Total: Total of all reporting groups
Arm/Group | Tucatinib+ Ado-trastuzumab Emtansine | Placebo+ Ado-trastuzumab Emtansine | Total
Number analyzed (Participants) | 228 | 235 | 463
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.8 (11.4) | 52.9 (10.9) | 53.4 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 226 | 235 | 461
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 13 | 21
  Not Hispanic or Latino | 171 | 163 | 334
  Unknown or Not Reported | 49 | 59 | 108
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 66 | 65 | 131
  Native Hawaiian or Other Pacific Islander | 3 | 0 | 3
  Black or African American | 11 | 8 | 19
  White | 101 | 102 | 203
  More than one race | 5 | 1 | 6
  Unknown or Not Reported | 42 | 58 | 100

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) as Per Response Evaluation Criteria in Solid Tumors (RECIST) Version (v)1.1 Based on Investigator Assessment
Description: PFS as per investigator was defined as the time from the date of randomization to the investigator assessment of disease progression (PD) as per RECIST v1.1 or death from any cause, whichever occurred first. PD: at least a 20 percent (%) increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimiter (mm). Participants without documentation of PD, or death at the time of analysis were censored at the date of the last tumor assessment.
Time Frame: From the date of randomization to the date of PD or death from any cause or censoring date, whichever occurred first (maximum up to 43 months)
Population: The ITT analysis set included all participants who were randomized on or before the date of LPI, in the global study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tucatinib+ Ado-trastuzumab Emtansine | Placebo+ Ado-trastuzumab Emtansine
Number analyzed (Participants) | 228 | 235
Months | 9.5 [7.4 to 10.9] | 7.4 [5.6 to 8.1]
Statistical Analysis 1: Comparison: Tucatinib+ Ado-trastuzumab Emtansine vs Placebo+ Ado-trastuzumab Emtansine; Test type: Other; p = 0.0163, Log Rank; Hazard Ratio (HR) = 0.759, 95% CI 2-sided [0.607 to 0.950] — HR was calculated from Cox proportional hazards model. (line of treatment for metastatic: first versus [vs] other; hormone receptor status: negative vs positive; presence or history of brain metastases: yes vs no; ECOG status: 0,1 at randomization

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause. For a participant who was not known to have died by the end of study follow-up, observation of OS was censored on the date the participant was last known to be alive (i.e., the date of last contact).
Time Frame: Up to approximately 5 years
Reporting Status: Not Posted, anticipated posting 2028-10

3. Secondary Outcome: Progression-Free Survival as Per RECIST v1.1 in Participants With Brain Metastases at Baseline Based on Investigator Assessment
Description: PFS as per investigator was defined as the time from the date of randomization to the investigator assessment of PD as per RECIST v1.1 or death from any cause, whichever occurred first. PD: at least a 20 % increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Participants without documentation of PD, or death at the time of analysis were censored at the date of the last tumor assessment. PFS was analyzed in participants with presence or history of brain metastases.
Time Frame: From the date of randomization to the date of PD or death from any cause or censoring date, whichever occurred first (maximum up to 45 months)
Population: The ITT analysis set included all participants who were randomized on or before the date of LPI, in the global study. Here "Overall Number of Participants Analyzed" signifies the number of participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tucatinib+ Ado-trastuzumab Emtansine | Placebo+ Ado-trastuzumab Emtansine
Number analyzed (Participants) | 99 | 105
Months | 7.8 [6.7 to 10.0] | 5.7 [4.6 to 7.5]
Statistical Analysis 1: Comparison: Tucatinib+ Ado-trastuzumab Emtansine vs Placebo+ Ado-trastuzumab Emtansine; Test type: Other; p = 0.0078, Log Rank; Hazard Ratio (HR) = 0.639, 95% CI 2-sided [0.459 to 0.891] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Objective Response Rate (ORR) as Per RECIST v1.1 Based on Investigator Assessment
Description: ORR was defined as the percentage of participants with confirmed complete response (CR) or partial response (PR) according to RECIST v1.1. CR: disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to less than (<)10 mm. PR: a greater than equal (>=) 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. For a response to be considered as confirmed, the subsequent response needs to be at least 4 weeks after the initial response. ORR by investigator assessment is based on investigator response assessments. Two-sided 95% exact confidence interval, computed using the Clopper-Pearson method.
Time Frame: From the date of first CR or PR until the date of the first documentation of PD or death, whichever occurred first (maximum up to 43 months)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tucatinib+ Ado-trastuzumab Emtansine | Placebo+ Ado-trastuzumab Emtansine
Number analyzed (Participants) | 188 | 191
Percentage of participants | 42.0 [34.9 to 49.4] | 36.1 [29.3 to 43.4]
Statistical Analysis 1: Comparison: Tucatinib+ Ado-trastuzumab Emtansine vs Placebo+ Ado-trastuzumab Emtansine; Test type: Other; p = 0.2055, Cochran-Mantel-Haenszel

5. Secondary Outcome: Overall Survival in Participants With Brain Metastases at Baseline
Description: OS was defined as the time from randomization to death due to any cause. For a participant who was not known to have died by the end of study follow-up, observation of OS was censored on the date the participant was last known to be alive (i.e., the date of last contact). OS was analyzed in participants with presence or history of brain metastases.
Time Frame: Up to approximately 5 years
Reporting Status: Not Posted, anticipated posting 2028-10

6. Secondary Outcome: Progression-Free Survival as Per RECIST v1.1 Determined by Blinded Independent Committee Review (BICR)
Description: PFS as per BICR was defined as the time from the date of randomization to the centrally-reviewed documented PD as per RECIST v1.1 or death from any cause, whichever occurred first. PD: at least a 20 % increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Participants without documented progression of PD or death at the time of analysis were censored at the date of the last tumor assessment.
Time Frame: as for outcome 1
Population: The ITT analysis set included all participants who were randomized on or before the date of LPI, in the global study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tucatinib+ Ado-trastuzumab Emtansine | Placebo+ Ado-trastuzumab Emtansine
Number analyzed (Participants) | 228 | 235
Months | 9.6 [7.5 to 10.9] | 7.4 [5.5 to 8.4]

7. Secondary Outcome: Progression-Free Survival in Participants With Brain Metastases at Baseline as Per RECIST v1.1 Determined by BICR
Description: PFS as per BICR was defined as the time from the date of randomization to the centrally-reviewed documented PD as per RECIST v1.1 or death from any cause, whichever occurred first. PD: at least a 20 % increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. PFS was analyzed in participants with presence or history of brain metastases.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tucatinib+ Ado-trastuzumab Emtansine | Placebo+ Ado-trastuzumab Emtansine
Number analyzed (Participants) | 99 | 105
Months | 7.8 [6.9 to 10.0] | 5.5 [4.2 to 7.4]

8. Secondary Outcome: Objective Response Rate as Per RECIST v1.1 Determined by BICR
Description: ORR was defined as the percentage of participants with confirmed CR or PR according to RECIST v1.1. CR: Disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm. PR: A >= 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. ORR per BICR is based on BICR response assessments.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tucatinib+ Ado-trastuzumab Emtansine | Placebo+ Ado-trastuzumab Emtansine
Number analyzed (Participants) | 182 | 185
Percentage of participants | 47.3 [39.8 to 54.8] | 41.1 [33.9 to 48.5]

9. Secondary Outcome: Duration of Response (DOR) as Per RECIST v1.1 Based on Investigator Assessment
Description: DOR was defined as the time from first documentation of objective response (CR or PR that is subsequently confirmed) to the first documentation of PD as per RECIST v1.1 PD: at least a 20 % increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Participants without documentation of PD, or death at the time of analysis were censored at the date of the last tumor assessment. CR: disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm. PR: A>=30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. DOR per investigator was based on investigator response assessments.
Time Frame: Up to approximately 5 years
Reporting Status: Not Posted, anticipated posting 2028-10

10. Secondary Outcome: Duration of Response as Per RECIST v1.1 by BICR
Description: DOR was defined as the time from first documentation of objective response (CR or PR that is subsequently confirmed) to the first documentation of PD as per RECIST v1.1 PD: at least a 20 % increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Participants without documentation of PD, or death at the time of analysis were censored at the date of the last tumor assessment. CR: disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm. PR: A>=30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. DOR per BICR was based on BICR response assessments.
Time Frame: Up to approximately 5 years
Reporting Status: Not Posted, anticipated posting 2028-10

11. Secondary Outcome: Clinical Benefit Rate (CBR) Per RECIST v1.1 Based on Investigator Assessment
Description: CBR was defined as the percentage of participants with stable disease (SD) or non-CR or non-PD >= 6 months or best response of CR or PR according to RECIST v1.1. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. CR: disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm. PR: A >= 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. CBR was based on investigator assessment.
Time Frame: Up to approximately 5 years
Reporting Status: Not Posted, anticipated posting 2028-10

12. Secondary Outcome: Clinical Benefit Rate as Per RECIST v1.1 by BICR
Description: CBR was defined as the percentage of participants with SD or non-CR or non-PD >= 6 months or best response of CR or PR according to RECIST v1.1. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. CR: disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm. PR: A >= 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. CBR per BICR is based on BICR response assessments.
Time Frame: Up to approximately 5 years
Reporting Status: Not Posted, anticipated posting 2028-10

13. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAE was defined as AE that is newly occurred or worsened after the start of study treatment.
Time Frame: From start of treatment up to 30 days after the last study treatment (approximately 43 months)
Population: The safety analysis set included all participants who were randomized or enrolled on or before the date of LPI in the global study and received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Tucatinib+ Ado-trastuzumab Emtansine | Placebo+ Ado-trastuzumab Emtansine
Number analyzed (Participants) | 231 | 233
Participants | 230 | 233

ADVERSE EVENTS:
Time Frame: From start of treatment up to 30 days after the last study treatment (approximately 43 months)
Description: Same event may appear as both non-serious adverse event (SAE) and SAE; however, what is presented are distinct events. An event may be categorized as serious in 1 participant and non-serious in other participant, or a participant may have experienced both SAE and non-SAE. The safety analysis set included all participants who were randomized or enrolled on or before the date of LPI in the global study and received at least 1 dose of study treatment.
Arm/Group | Placebo+ Ado-trastuzumab Emtansine | Tucatinib+ Ado-trastuzumab Emtansine
All-Cause Mortality (participants affected / at risk) | 63/233 | 71/231
Serious Adverse Events (participants affected / at risk) | 52/233 | 70/231
Other Adverse Events (participants affected / at risk) | 227/233 | 230/231
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo+ Ado-trastuzumab Emtansine (N=233) | Tucatinib+ Ado-trastuzumab Emtansine (N=231)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 1 (1)
Otorrhoea (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 3 (3)
Chest pain (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (3) | 1 (1)
Gait inability (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 3 (3)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 2 (3)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 3 (3)
Hepatic failure (Hepatobiliary disorders) | 2 (2) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 2 (2)
Cellulitis (Infections and infestations) | 1 (2) | 1 (1)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (2)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Mastitis (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 4 (4) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia fungal (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 4 (5) | 4 (4)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 2 (2)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Brain herniation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Splenic injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Ejection fraction decreased (Investigations) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hyperammonaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 2 (2) | 2 (2)
Central nervous system necrosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 1 (3) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 2 (2) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Post herpetic neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 3 (3) | 3 (4)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (3) | 3 (3)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo+ Ado-trastuzumab Emtansine (N=233) | Tucatinib+ Ado-trastuzumab Emtansine (N=231)
Anaemia (Blood and lymphatic system disorders) | 26 (35) | 44 (58)
Thrombocytopenia (Blood and lymphatic system disorders) | 29 (33) | 37 (44)
Dry eye (Eye disorders) | 14 (14) | 24 (26)
Vision blurred (Eye disorders) | 23 (27) | 23 (25)
Abdominal pain (Gastrointestinal disorders) | 28 (33) | 34 (40)
Abdominal pain upper (Gastrointestinal disorders) | 21 (30) | 25 (33)
Constipation (Gastrointestinal disorders) | 77 (99) | 61 (76)
Diarrhoea (Gastrointestinal disorders) | 62 (92) | 131 (217)
Dry mouth (Gastrointestinal disorders) | 31 (31) | 25 (25)
Dyspepsia (Gastrointestinal disorders) | 23 (26) | 24 (28)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 16 (17)
Gingival bleeding (Gastrointestinal disorders) | 12 (13) | 7 (9)
Nausea (Gastrointestinal disorders) | 113 (152) | 151 (260)
Stomatitis (Gastrointestinal disorders) | 31 (41) | 16 (16)
Vomiting (Gastrointestinal disorders) | 39 (59) | 85 (153)
Asthenia (General disorders) | 31 (55) | 28 (39)
Chills (General disorders) | 12 (13) | 17 (26)
Fatigue (General disorders) | 85 (115) | 113 (151)
Malaise (General disorders) | 10 (22) | 12 (14)
Oedema peripheral (General disorders) | 18 (22) | 20 (24)
Pain (General disorders) | 5 (5) | 12 (15)
Pyrexia (General disorders) | 33 (43) | 54 (94)
COVID-19 (Infections and infestations) | 35 (39) | 37 (39)
Nasopharyngitis (Infections and infestations) | 15 (16) | 10 (12)
Upper respiratory tract infection (Infections and infestations) | 12 (13) | 8 (8)
Urinary tract infection (Infections and infestations) | 21 (27) | 29 (52)
Contusion (Injury, poisoning and procedural complications) | 10 (10) | 16 (21)
Fall (Injury, poisoning and procedural complications) | 11 (13) | 15 (23)
Infusion related reaction (Injury, poisoning and procedural complications) | 6 (7) | 15 (18)
Alanine aminotransferase increased (Investigations) | 40 (56) | 78 (103)
Aspartate aminotransferase increased (Investigations) | 45 (61) | 83 (115)
Blood alkaline phosphatase increased (Investigations) | 6 (7) | 12 (17)
Blood bilirubin increased (Investigations) | 14 (27) | 27 (72)
Platelet count decreased (Investigations) | 20 (27) | 25 (46)
Weight decreased (Investigations) | 14 (15) | 34 (34)
Decreased appetite (Metabolism and nutrition disorders) | 53 (65) | 78 (99)
Dehydration (Metabolism and nutrition disorders) | 8 (8) | 16 (18)
Hypokalaemia (Metabolism and nutrition disorders) | 25 (33) | 32 (39)
Hypomagnesaemia (Metabolism and nutrition disorders) | 11 (17) | 13 (18)
Arthralgia (Musculoskeletal and connective tissue disorders) | 63 (88) | 54 (75)
Back pain (Musculoskeletal and connective tissue disorders) | 35 (43) | 25 (26)
Bone pain (Musculoskeletal and connective tissue disorders) | 8 (12) | 13 (15)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 17 (18) | 25 (28)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 9 (10) | 12 (12)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 12 (12) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 29 (32) | 37 (37)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 29 (44) | 27 (33)
Dizziness (Nervous system disorders) | 30 (33) | 30 (32)
Dysgeusia (Nervous system disorders) | 14 (14) | 16 (20)
Headache (Nervous system disorders) | 90 (131) | 83 (120)
Peripheral sensory neuropathy (Nervous system disorders) | 47 (62) | 41 (43)
Anxiety (Psychiatric disorders) | 13 (13) | 17 (17)
Depression (Psychiatric disorders) | 7 (7) | 12 (12)
Insomnia (Psychiatric disorders) | 28 (30) | 28 (32)
Cough (Respiratory, thoracic and mediastinal disorders) | 38 (48) | 38 (43)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23 (27) | 25 (28)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 46 (63) | 79 (125)
Dry skin (Skin and subcutaneous tissue disorders) | 18 (18) | 23 (23)
Pruritus (Skin and subcutaneous tissue disorders) | 19 (21) | 18 (24)
Rash (Skin and subcutaneous tissue disorders) | 17 (23) | 32 (35)
Rash macular (Skin and subcutaneous tissue disorders) | 7 (7) | 12 (21)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 18 (23) | 23 (30)
Hypertension (Vascular disorders) | 8 (13) | 14 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-11-08): https://cdn.clinicaltrials.gov/large-docs/47/NCT03975647/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-31): https://cdn.clinicaltrials.gov/large-docs/47/NCT03975647/SAP_001.pdf